CLINICAL TRIAL: NCT04159493
Title: A Randomized, Double-blind, Placebo-Controlled, Dose De-escalation Phase 2 Study of Various Doses of Ovestin in the Treatment of Symptoms of Vulvar and Vaginal Atrophy in Postmenopausal Women
Brief Title: A Randomized Controlled Phase 2 Study to Determine Lowest Efficacious Dose of Ovestin in Vulvar and Vaginal Atrophy
Acronym: DOVE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Project terminated IND withdrawn
Sponsor: Aspen USA Inc (Industry)
Responsible Party: Sponsor
Organization: Aspen Global Incorporated (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLINTECUS-19-OVDFP2
Record Dates: First submitted 2019-10-22; First posted 2019-11-12 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Vaginal Atrophy
MeSH Terms: interventions — Estriol

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, randomized, double-blind, placebo-controlled, dose de-escalation study whose purpose is to establish the lowest efficacious dose of Ovestin
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be randomized to placebo.
  Placebo, Vaginal Application 0.5 to 2 g administered daily for the 1st 14 days, then twice weekly for following 10 weeks
  Interventions: Drug: Placebo
- Ovestin (Active Comparator): Subjects will be randomized or assigned to varying doses of Ovestin (500, 50, 25, 12.5, 10, 5, 2.5, 0.5, 0.25 mcg) as determined by the dose de-escalation constraints specified in the protocol.
  Active, Vaginal Application 0.5 to 2 g administered daily for the 1st 14 days, then twice weekly for following 10 weeks
  Interventions: Drug: Estriol

INTERVENTIONS:
Drug: Estriol — Vaginal Application
  Other Names: Ovestin
  Arms: Ovestin
Drug: Placebo — Vaginal Application
  Arms: Placebo

SUMMARY:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled, dose-de-escalation study whose purpose is to establish the lowest efficacious dose. The first 40 subjects will be randomized 1:1:1:1 to either 500 mcg, 50 mcg, 10 mcg, or placebo. After four weeks of dosing with 500 mcg, vaginal pH, vaginal maturation index, and subject's most bothersome moderate to severe symptom will be assessed; the changes observed will be used as the benchmark for efficacy throughout the remainder of the study and select the next dose-level to be investigated. Subjects will be enrolled in small cohorts at various doses until the lowest effective dose is identified. Then, 1 to 2 doses and a placebo group will be expanded to enroll 70 subjects per treatment group.

DETAILED DESCRIPTION:
For each dose, an initial efficacy determination will be made based on changes in vaginal pH, vaginal maturation index, and patient's most bothersome moderate to severe symptom after four weeks of dosing. Depending on the initial efficacy results, one of the following dosing schemes may occur:

* If 50 mcg is determined to be inefficacious, 10 additional subjects will be enrolled at 50 mcg. If 50 mcg is now determined to be efficacious, the dosing cohort will be expanded to 70 subjects at 50 mcg. If 50mcg is determined to be inefficacious, no groups will be expanded to 70 subjects.
* If 10 mcg is determined to be efficacious, an additional 10 subjects will be enrolled to 2.5 mcg. If 2.5 mcg is determined to be efficacious, 10 subjects will be enrolled to 0.25 mcg. If 0.25 mcg is efficacious, 0.25 mcg and 0.5 mcg will be enrolled to a total of 70 subjects per dose. If 0.25 mcg is determined to be inefficacious, 10 subjects will be enrolled to 0.5 mcg. If 0.5 mcg is determined to be efficacious, 0.5 mcg and 2.5 mcg will be enrolled to 70 subjects per dose. If 0.5 mcg is determined to be inefficacious, 2.5 mcg and 5 mcg will be enrolled to 70 subjects per dose. If 2.5 mcg is determined to be inefficacious, 10 subjects will be enrolled to 5 mcg. If 5 mcg is determined to be efficacious, 5 mcg and 10 mcg will be enrolled to 70 subjects per dose. If 5 mcg is determined to be inefficacious, 10 mcg and 12.5 mcg will be enrolled to 70 subjects per dose.
* If 10 mcg is determined to be inefficacious, 10 subjects will be enrolled to 25 mcg. If 25 mcg is determined to be efficacious, 10 subjects will be enrolled to 12.5 mcg. If 12.5 mcg is determined to be efficacious, 12.5 mcg and 25 mcg will be enrolled to 70 subjects per dose. If 12.5 mcg is determined to be inefficacious, 25 mcg and 50 mcg will be enrolled to 70 subjects per dose. If 25 mcg is inefficacious, 50 mcg will be expanded to 70 subjects.

Subjects will be randomized 1:1:1 for each of the two doses selected and placebo for expansion to 70 subjects. For all doses evaluated, the mean change from baseline in vaginal maturation index and vaginal pH and the mean change from baseline in the most bothersome symptom will be assessed at the end of 12 weeks.

Evaluation After 4 weeks of Dosing After four weeks of dosing, each dose will be assessed for its efficaciousness in altering the vaginal maturation index, the vaginal pH, and the most bothersome moderate to severe symptom. The response identified in the subjects dosed in the 500 mcg cohort relative to placebo at four weeks will serve as the effect of the active control to assess the efficaciousness of the other dose levels. After reviewing these results, the sponsor will determine the assessment of subsequent dose levels.

ELIGIBILITY:
Subjects must meet the following criteria to be included in the study:

1. Body mass index (BMI) between 18 and 38 kg/m2
2. Presence of at least one documented moderate or severe bothersome symptom of vulvovaginal atrophy. These symptoms include either:

   1. Vaginal dryness
   2. Vaginal itching/irritation

5. Postmenopausal women; postmenopausal defined as:

a. 12 months of spontaneous amenorrhea, or b. 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy c. 6-12 months of spontaneous amenorrhea with serum follicle stimulating (FSH) levels of > 40 mIU/mL. 3. Participants will comprise treatment-naïve postmenopausal women and treatment-experienced postmenopausal women who have discontinued hormone replacement therapy (either local or systemic) 4. Participants should not be taking estrogen alone or estrogen/progestin containing drug products. The following washout periods are recommended before baseline assessments are made for participants previously on estrogen alone or estrogen/progestin containing products:

1. 4 weeks or longer for prior vaginal hormonal products (rings, creams, gels)
2. 4 weeks or longer for prior transdermal estrogen alone or estrogen/progestin products
3. 8 weeks or longer for prior oral estrogen and/or progestin therapy
4. 8 weeks or longer for prior intrauterine progestin therapy
5. 3 months or longer for prior progestin implants and estrogen alone injectable drug therapy
6. 6 months or longer for prior estrogen pellet therapy or progestin injectable drug therapy 5. Participants must agree to refrain from use of any water-based or oil-based vaginally administered products (e.g. vaginal antifungal products or vaginal lubricants) throughout the study, a 5-day washout will apply.

   6. Women must have documentation of a negative screening mammogram (obtained at screening or within nine months prior to study enrollment) and normal clinical breast examination prior to enrollment.

   7. Women must have documentation of a negative screening pap smear (obtained at screening or within six months prior to study enrollment). Negative defined as normal cytology or pap1 (normal cytomorphology) or pap2 (borderline dyskaryosis/ atypical squamous cells of undetermined significance (ASC-US) and no suspected malignant abnormalities.

   8. Participants must sign an informed consent consistent with ICH-GCP guidelines prior to participation in the trial.

   9. Women must have a documented negative urine pregnancy test unless they have had a bilateral oophorectomy and/or hysterectomy.

   10. Women must have a 5% superficial epithelial cells on a lateral wall vaginal smear.

   11. Women must have a vaginal pH >5. 12. Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria

Subjects will be excluded from the study for:

1. History of endometrial hyperplasia or cervical cancer for participants who have a uterus.
2. Known, previous or suspected breast cancer.
3. Known, previous or suspected estrogen-dependent malignant tumors (e.g. endometrial cancer). In participants with a uterus, the histological diagnosis of disordered proliferative endometrium, endometrial hyperplasia or cancer based on endometrial biopsy.
4. Any malignancy unless free of disease for at least 5 years.
5. Know hypersensitivity to the active substance or any of the excipients.
6. Undiagnosed uterine bleeding.
7. Known pelvic organ prolapse past the level of the hymen.
8. Evidence of vaginal infection on physical examination.
9. Previous or current venous thromboembolism (deep venous thrombosis, pulmonary embolism).
10. Active or recent arterial thromboembolic disease (e.g. angina or myocardial infarction)
11. Known thrombophilic disorders or conditions that may adversely affect coagulation, including:

    1. Protein C, Protein S, or antithrombin III deficiency
    2. Factor XIII mutation, dysfibrinogenemia, antiphospholipid syndrome, heparin-induced thrombocytopenia, paroxysmal nocturnal hemoglobinuria, sickle-cell disease, polycythemia vera, essential thrombocytosis, nephrotic syndrome
    3. History of elevated levels of factor VIII, factor IX, factor XI, fibrinogen and thrombin-activatable fibrinolysis inhibitor, or decreased levels of tissue factor pathway inhibitor
12. Acute or chronic liver disease.
13. Subjects with hypertension defined as systolic blood pressure >140 mmHg and/or diastolic blood pressure > 90 mmHg are excluded based on an average of two or three readings on at least two different occasions. Subjects with systolic blood pressure >130 mmHg or diastolic blood pressure >80 mmHg, based on an average of two to three readings on at least two different occasions, may be enrolled if cleared by a physician.
14. A history of significant alcohol or drug abuse in the opinion of the investigator.
15. Use of any other investigational drug within 30 days or use of any of the prohibited medications, leading up to the first dose of Ovestin.
16. Any physical, psychiatric or social condition which in the opinion of the investigator may:

    1. Put the participant at risk because of participation in the study
    2. Influence the results of the study
    3. Cause concern regarding the participant's ability to participate in the study

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Post-menopausal women aged 45 to 85 years at randomization will be enrolled to the study.
Enrollment: 0 (Actual)
Dates: Start 2021-06-05 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Vaginal Maturation Index | 12 weeks
  Mean change from baseline at Week 12 in vaginal maturation index (percentage of superficial and parabasal cells)
Vaginal pH | 12 Weeks
  Mean change from baseline at Week 12 in vaginal pH
Most Bothersome Symptom | 12 weeks
  Mean change from baseline at Week 12 in the moderate to severe symptom that has been identified by the subject as being the most bothersome to her

SECONDARY OUTCOMES:
Incidence of adverse events | 12 weeks
  To evaluate the safety profile of Ovestin at doses evaluated

IPD SHARING:
Plan to Share IPD: No